CLINICAL TRIAL: NCT02652078
Title: Extracorporeal Shockwave Therapy in the Treatment of Intermittent Claudication Symptoms in Peripheral Vascular Disease
Brief Title: Shockwave Therapy in Lower Limb Intermittent Calf Claudication
Acronym: ESWT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shockwave 1; 166137 (Other: IRAS project ID)
Record Dates: First submitted 2014-10-17; First posted 2016-01-11 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Sham treatment in identical format to treatment arm but without shockwave production
  Interventions: Device: Extracorporeal shockwave therapy
- Shockwave (Experimental): Active shockwave treatment to calf muscle bulk
  Interventions: Device: Extracorporeal shockwave therapy

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — Ultrasonic shockwaves targeted at calf muscle bulk using the Piezowave 2 device (Richard Wolf, Knittlingen, Germany)
  Other Names: external shockwave

SUMMARY:
Peripheral arterial disease is a common condition affecting approximately 64% of 56-77 year olds. This condition restricts bloody supply to calf muscles. Pain occurs after walking a short distance and increases in intensity until the person stops, where the pain then gradually subsides. It can be limiting or occasionally debilitating and has been shown to have considerable deleterious effects of patients quality of life. Shock wave therapy has been shown to promote new blood vessel formation and improved healing amongst other findings. This study aims to identify whether shock wave therapy that is applied to the calf muscles causes such an effect to improve the blood supply to the calf muscles, reduce pain, improve walking ability and quality of life.

DETAILED DESCRIPTION:
This study aims to compare the effects of extracorporeal shockwave therapy (ESWT) to placebo with use of a sham control group on walking distances in subjects with lower limb intermittent calf claudication. Extracorporeal shockwave therapy will be applied using the PiezoWave2 shockwave system. All applications will be in adherence to the manufacturer's instructions and provided by trained staff. The device will be targeted at the gastrocnemius muscles of the affected lower leg for several minutes at each treatment session. Participants in control group will undergo the identical process as if treatment were being given but with the shockwaves not being administered and a sham device alternatively used. Participants will have several assessments prior to and after the shockwave treatment in order to quantify the effect. Assessments will include Maximum Walking Distance (MWD), Claudication Distance (CD) and Quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral intermittent calf claudication (stable for the last 3 months).
* Able to give written informed consent to participate in the study
* Age > 18
* Able to adhere to protocol and attend all follow up appointments
* Currently receiving "best medical therapy" - anti-platelet and statin medication

Exclusion Criteria:

* Current malignancy
* Allergies or intolerances of either anti-platelet medication or statin therapy
* Pregnancy (pregnancy test performed at screening if necessary)
* Metal implant near to treatment area
* Anti-coagulation medication (i.e. Warfarin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Walking Distance (MWD) | 12 weeks
  Treadmill test

SECONDARY OUTCOMES:
Claudication Distance | 12 weeks
  Distance covered prior to onset of any symptoms
Changes in Ankle Brachial Pressure Index | Week 4, 8 and 12
Changes in Patient reported walking distance | Week 4, 8 and 12
Changes in Quality of life [Short form 36(SF36) | Week 4, 8 and 12
Changes in Quality of life [EuroQoL (EQ5D)] | Week 4, 8 and 12
Subject tolerance of treatment | Week 4
  Questionnaire including visual analogue pain scales

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chetter, Principal Investigator — Hull and East Yorkshire Hospital Trust
Locations (1):
- Academic Vascular Surgery Unit, Hull, Yorkshire, United Kingdom

REFERENCES:
- [Result] Green JL, Harwood AE, Smith GE, Das T, Raza A, Cayton T, Wallace T, Carradice D, Chetter IC. Extracorporeal shockwave therapy for intermittent claudication: Medium-term outcomes from a double-blind randomised placebo-controlled pilot trial. Vascular. 2018 Oct;26(5):531-539. doi: 10.1177/1708538118773618. Epub 2018 May 3. PMID 29722640
- [Result] Cai P, Pymer S, Ibeggazene S, Raza A, Hitchman L, Chetter I, Smith G. Extracorporeal Shockwave for Intermittent Claudication and Quality of Life: A Randomized Clinical Trial. JAMA Surg. 2024 Jun 1;159(6):625-632. doi: 10.1001/jamasurg.2024.0625. PMID 38598227
- [Derived] Harwood AE, Green J, Cayton T, Raza A, Wallace T, Carradice D, Chetter IC, Smith GE. A feasibility double-blind randomized placebo-controlled trial of extracorporeal shockwave therapy as a novel treatment for intermittent claudication. J Vasc Surg. 2018 Feb;67(2):514-521.e2. doi: 10.1016/j.jvs.2017.07.105. Epub 2017 Sep 22. PMID 28943002
- [Derived] Cayton T, Harwood AE, Smith GE, Totty JP, Carradice D, Chetter IC. Extracorporeal shockwave therapy for the treatment of lower limb intermittent claudication: study protocol for a randomised controlled trial (the SHOCKWAVE 1 trial). Trials. 2017 Mar 6;18(1):104. doi: 10.1186/s13063-017-1844-4. PMID 28264725
- See also: Publication Link — https://www.ncbi.nlm.nih.gov/pubmed/29722640?dopt=Abstract